CLINICAL TRIAL: NCT00365534
Title: A Double-Blinded Randomized Study Comparison the Mechanism of Looping Formation and Subject's Acceptance During CAC and Regular Colonoscopy by MEI (MIC Study)
Brief Title: Use of Magnetic Imaging to Asses the Efficacy of Cap Assisted Colonoscopy in Reducing Looping and Improving Patient Acceptance for the Colonoscopy Procedure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was incorporated in another study.
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: MIC
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Colonoscopy
Keywords: First colonoscopy examination

INTERVENTIONS:
Procedure: MEI

SUMMARY:
The aim of this study is to compare the mechanism of loop formation and acceptance of CAC and regular colonoscopy by MEI.

DETAILED DESCRIPTION:
Colonoscopy is widely used for the investigation of lower gastrointestinal tract disease.However,colonoscopy remains a technically difficult procedure. As the colon is a mobile organ, looping may occur when the colonoscope passes through.Hence,reducing looping during procedure is very improtant to achieve succes as well as patient acceptance.Recently,some studies shown that cap-assisted colonoscopy(CAC)allow better visualisation of the colonic folds, thus increase success rate.However, previous studies shown that magnetic endoscope imaging (MEI)is useful as an adjunct to assist endoscopist in performing the procedure and as a modality to look for the mechanism of looping. Because of such concern,our study is to compare the mechanism of looping formation and acceptance of CAC and regular colonoscopy by MEI.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergo first colonoscopy examination
* Signed informed consent

Exclusion Criteria:

* Patient had received colonoscopy examination before.
* Patient had prior colorectal surgery done(apart from appendectomy)
* Known to have colonic stricture or obstructing tumour from the result of other investigations such as CT scan or barium enema.
* Presence of acute surgical conditions such as severe colitis, megacolon, ischaemic colitis and active gastrointestinal bleeding.
* Patient could not provide consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01

PRIMARY OUTCOMES:
The MEI score difference between regular colonoscopy and CAC.

CONTACTS AND LOCATIONS:
Overall Officials: Yuk Tong Lee, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre,Alice Ho Miu Ling Nethersole Hospital & Tai Po Hospital, Hong Kong, China